CLINICAL TRIAL: NCT02740881
Title: Online Training Support System for Community-Based Substance Abuse Agencies
Brief Title: Web-Based Contingency Management Training for Addictions
Acronym: CM-TSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheidow Consulting, Inc. (Other)
Collaborators: Oregon Social Learning Center (Other)
Responsible Party: Principal Investigator, Jaime Mulligan, Vice President, Sheidow Consulting, Inc.
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: R44DA033745 (NIH)
Record Dates: First submitted 2015-11-25; First posted 2016-04-15 (Estimated); Last update posted 2018-12-31 (Actual); Status verified 2018-12

CONDITIONS: Substance Abuse Problem
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Training Support System (Experimental): Participants receive training in Contingency Management and immediately receive the full training support system and quality assurance feedback for 15 months while they provide the treatment.
  Interventions: Other: Counselor Training Methods
- CM-CAT then TSS (Active Comparator): Participants are trained in Contingency Management and use the treatment without training support and quality assurance feedback for 9 months. After 9 months they continue using Contingency Management but now receive the full training support system and quality assurance feedback for 6 months.
  Interventions: Other: Counselor Training Methods

INTERVENTIONS:
Other: Counselor Training Methods

SUMMARY:
Adolescent substance abuse results in significant negative outcomes and extraordinary costs for youths, their families, communities and society (societal costs estimated at over $400 billion annually and greater than costs for any other health problem). There is a clear public health need for improving and expanding the delivery of evidence-based treatments for adolescent substance use, but despite this clear need, there is a large divide between science and practice. This project will develop a cost-effective, easily accessible, web-based Training Support System (TSS) for Contingency Management that incorporates ongoing training, feedback, and support provided to both counselors and their community-based agencies.

DETAILED DESCRIPTION:
Drug abusing and dependent youth represent a greatly under-served population at high risk of presenting significant deleterious long-term outcomes for themselves, their families, communities and society at extraordinary long-term costs. Adolescent substance use has been linked to serious problems including automobile accidents, increased rates of risky sexual behavior which increases the youth's chances of contracting sexually transmitted diseases, high rates of physical and sexual abuse, and increased risk for school dropout. Further, drug use during adolescence predicts decreased college involvement as well as direct links to unemployment and job instability in young adulthood. In general, youth with substance use disorders represent a greatly under-served population in need of effective treatment; however, adolescents and their families seeking treatment are unlikely to receive an effective evidence-based intervention. Given this, there is a clear public health need for improving and expanding the delivery of evidence-based treatments for adolescent substance use. Despite this clear need, there is a large divide between science and practice. The proposed project has the potential to overcome a gaping need within the outpatient treatment sector, which is the largest purveyor of adolescent substance use treatment in the country. Specifically, the proposed SBIR Phase II project will commercialize a targeted internet-based Training Support System (TSS) which will make it possible for community-based agencies to adopt, implement, and sustain use of Contingency Management (CM), an evidence-based substance abuse treatment for adolescents and their families. This system includes an initial computer assisted training for individual counselors, individual- and agency-level performance assessment and feedback processes, remediation training and support, organizational-level consultation on funding structures, and clinical expert guidance for counselors. This entirely internet-based training and support system is the first of its kind. It provides a cost-effective training and support platform for community-based substance abuse treatment providers, enabling them to train staff in an evidence-based practice with the necessary ongoing support to ensure fidelity and rapid uptake of the practice. The Phase I aims focused on development of the TSS and initial pilot testing. The Phase II project's first aim is to finalize development of the TSS based on data collected in the Phase I pilot testing. These data-driven enhancements and changes will ensure high usability and commercialization potential of the TSS. The project's second aim is to conduct a randomized trial evaluating the efficacy of the TSS in community-based settings, including qualitative evaluation of the TSS and quantitative evaluation of (a) counselor knowledge, adherence, and satisfaction and (b) clinical outcomes and client satisfaction. Phase II will conclude with the development of a market-ready CM Training Support System for community-based counselors that will provide a cost-effective strategy for increasing the use of evidence-based interventions for youth who need them and rarely have access to them.

ELIGIBILITY:
Inclusion Criteria:

* Professional counselors in outpatient substance abuse treatment agencies.
* Must treat adolescent substance abusers in clinic-based care.
* Counselors employed by these agencies are healthy, gainfully-employed individuals who are all adults with advanced degrees.

Exclusion Criteria:

* Participants will be excluded if they are not professional counselors
* Younger than age 22
* Do not work in outpatient substance abuse treatment agencies.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2015-11; Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Impact of training support on outpatient counselor fidelity to Contingency Management Substance Abuse Treatment Model measured using CM Therapist Adherence Measure (CM-TAM) | 15 months
  Impact of ongoing training and support on counselor fidelity to the Contingency Management treatment model will be measured through the administration of the Contingency Management Therapist Adherence Measure (CM-TAM), a 34 item paper and pencil survey, completed monthly through the duration of the study. Scores on the CM-TAM indicate amount of counselor adherence to the treatment model.
Impact of training support on outpatient counselor fidelity to Contingency Management Substance Abuse Treatment Model measured using session tape review and scoring | 15 Months
  Impact of ongoing training and support on counselor fidelity to the Contingency Management treatment model will be measured through the review and scoring of session audio tapes. Scores generated through the session tape review indicate amount of counselor adherence to the treatment model and extent of treatment implementation.
Impact of training support on outpatient counselor knowledge of, and fidelity to, the Contingency Management Substance Abuse Treatment Model measured using Contingency Management Knowledge Test (CM-KT) | 15 Months
  Impact of ongoing training and support on counselor fidelity to the Contingency Management treatment model will be measured through the administration of the Contingency Management Knowledge Test (CM-KT), a brief multiple choice tests administered annually. Scores from the CM-KT administrations summarize counselor knowledge changes over time.
Impact of training support on outpatient counselor fidelity to Contingency Management Substance Abuse Treatment Model measured using treatment outcomes. | 15 Months
  Impact of ongoing training and support on counselor fidelity to the Contingency Management treatment model and on treatment outcomes will be measured through the review of treatment outcomes.
Impact of training support on client satisfaction with treatment. | 15 months
  Impact of training support on client satisfaction with treatment will be measured using the Client Satisfaction Questionnaire (CSQ-8), completed by each client at the end of treatment.
Assessment of Counselor Training Satisfaction with Satisfaction Survey administration. | 15 months
  Counselor satisfaction with the training and training support will be measured using a counselor training satisfaction questionnaire. Counselors will complete 3 training satisfaction surveys over the course of the study.
Assessment of Counselor Satisfaction with Training and Training Support with Focus Group Outcomes | 15 months
  Counselor will participate in 2-3 focus groups (depending on condition assignment) over the course of the study. Focus groups will be used to gather qualitative information about the counselor experience with the training and support strategies.

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Mulligan, Psy.D., Principal Investigator — Sheidow Consulting, Inc.
Locations (1):
- Sheidow Consulting, Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: No